CLINICAL TRIAL: NCT03899974
Title: Metabolic Effects of High-amylose Wheat-based Breads in Overweight Individuals
Brief Title: Metabolic Effects of High-amylose Wheat-based Breads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 252/17
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 70% amylose bread (Experimental): Mixed meal with 80g of available carbohydrates coming mainly from high-amylose bread (made with 70% high-amylose flour)
  Interventions: Other: Test meal
- 85% amylose bread (Experimental): Mixed meal with 80g of available carbohydrates coming mainly from high-amylose bread (made with 85% high-amylose flour)
  Interventions: Other: Test meal
- Control bread (Active Comparator): Mixed meal with 80g of available carbohydrates coming mainly from conventional bread
  Interventions: Other: Test meal

INTERVENTIONS:
Other: Test meal — Participants received in random order the three test meal (700Kcal, 80g available carbohydrates) containing breads prepared with amylose-rich wheat flours (70% or 85%) or conventional flour. Blood samples were collected at fasting and every 30 minutes over 4 hours. Breath hydrogen was evaluated as a marker of intestinal fermentation. Participants underwent Visual Analogue Scale to assess subjective appetite sensations.
  After 4 hours, all participants consumed a standard lunch (700 kcal, 100 g available carbohydrates) identical on all the three experimental days to evaluate the "second meal effect" from breakfast to lunch.

SUMMARY:
The amylose-amylopectin ratio influences starch properties. A higher amylose content is associated with slower starch digestion thus reducing the postprandial plasma glucose response and improving the overall postprandial metabolism. So far, limited evidence is available on the metabolic effect of wheat-based foods rich in amylose. This randomised controlled study investigated the acute metabolic effects of amylose-rich wheat-based breads in overweight subjects focusing on potential mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese
* 18-70 years

Exclusion Criteria:

* age <18 and >70 years;
* fasting triglycerides ≥400 mg/dl;
* fasting cholesterol >270 mg/dl;
* cardiovascular events (myocardial infarction or stroke) during the 6 months prior to the study
* established diabetes mellitus or any chronic disease
* renal and liver failure (creatinine >1.7 mg/dl and transaminases >2 times than normal values, respectively)
* anaemia (Hb <12 g /dl)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
2-hours blood glucose response | over 2 hours after the test meal
  incremental area under the curve

SECONDARY OUTCOMES:
2-hours blood insulin response | over 2 hours after the test meal
  incremental area under the curve
4-hours blood glucose response | over 4 hours after the test meal
  incremental area under the curve
4-hours blood insulin response | over 4 hours after the test meal
  incremental area under the curve
intestinal fermentation | over 4 hours after the test meal
  breath test for the detection of hydrogen production
glucose response | over 2 hours after the standard meal
  Second meal effect

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Napoli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costabile G, Vetrani C, Calabrese I, Vitale M, Cipriano P, Salamone D, Testa R, Paparo L, Russo R, Rivellese AA, Giacco R, Riccardi G. High Amylose Wheat Bread at Breakfast Increases Plasma Propionate Concentrations and Reduces the Postprandial Insulin Response to the Following Meal in Overweight Adults. J Nutr. 2023 Jan;153(1):131-137. doi: 10.1016/j.tjnut.2022.10.007. Epub 2022 Dec 20. PMID 36913446